CLINICAL TRIAL: NCT00875537
Title: Neurogenic Mechanisms in Burning Mouth Syndrome With Focus on Localization and Desensibilization of Vanilloid Receptor TRPV1
Brief Title: Neurogenic Mechanisms in Burning Mouth Syndrome
Acronym: BMS17
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anne Marie Lynge Pedersen, Associate Professor, PhD, DDS, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-A-2008-118
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Burning Mouth Syndrome
Keywords: Burning mouth syndrome; neuropathy; inflammation; tongue mucosa; tongue innervation; dysgeusia
MeSH Terms: conditions — Burning Mouth Syndrome; Inflammation; Dysgeusia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capsaicin oral gel 0.01% (Active Comparator)
  Interventions: Other: Capsaicin oral gel 0.01%
- Capsaicin oral gel 0.025% (Active Comparator)
  Interventions: Other: Capsaicin oral gel 0.025%

INTERVENTIONS:
Other: Capsaicin oral gel 0.025% — Application 3 times daily for 14 days on the tongue, followed by 14 days wash-out
  Other Names: Capsicum, extract from chilipepper
  Arms: Capsaicin oral gel 0.025%
Other: Capsaicin oral gel 0.01% — Application 3 times daily for 14 days on the tongue, followed by 14 days wash-out
  Other Names: Capsicum, extract from chilipepper
  Arms: Capsaicin oral gel 0.01%

SUMMARY:
Burning mouth syndrome (BMS) is characterized by a bilateral burning sensation in the anterior tongue, hard palate and lips in the absence of any clinical or laboratory findings. The term syndrome implicates the simultaneous presence of oral dryness (xerostomia) and altered taste (dysgeusia) in addition to the burning sensation in the oral mucosa. BMS is most often seen in women and is more frequent during menopause. The etiology and pathogenesis are still unclear but recent studies suggest that BMS is a neuropathic pain condition.

The objectives of the study are:

* To clarify potential neurogenic mechanisms behind BMS using immunohistochemistry (IH) to characterize the localization and distribution of peripheral nerve fibres, neuropeptides like substance P, calcitonin gene-related peptide, nerve growth factor, nerve growth factor receptor, PGP 9.5 neuronal marker and TRPV1 as well as inflammatory/structural changes.
* To perform a randomized double blind cross-over intervention study to examine the efficacy and safety of topical application of capsaicin oral gel (on the tongue) to relieve the burning sensation in patients with BMS.

DETAILED DESCRIPTION:
Data which support the hypothesis that BMS is a neuropathic pain condition include amongst others a recent clinically controlled study that has shown up-regulation of TRPV1-positive nerve fibres in tongue mucosa in patients with BMS. The vanilloid receptor-1 (TRPV1) is a voltage-dependent cation channel expressed by the unmyelinated C-nociceptive nerve fibres and the receptor may be activated by capsaicin (from chili peppers), heat and H+. Capsaicin binds to the TRPV1 receptor causing depolarization of the C-nociceptors. Prolonged activation of these neurons by capsaicin depletes pre-synaptic substance P and makes them unable to report pain.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking female patients with burning mouth syndrome (n=26)
* healthy aged-matched control group (n=10)

Exclusion Criteria:

* pregnancy and lactation (inclusion requires negative pregnancy test)
* women who do not use safe anticonception
* patients with know allergy/hypersensitivity to capsicum and other capsaicinoid-containing products
* Active infection which requires antibiotic treatment
* use of mouthrinse. The use of these is stopped 14 days before inclusion
* patients who are able to give informed consent due to physical or mental disabilities

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome: To evaluate the efficacy and safety of topical application of capsaicin oral gel (using to different concentrations) to relieve the burning sensation in patients with BMS and alleviate BMS related symptoms. | 6 months

SECONDARY OUTCOMES:
To characterize the localization and distribution of peripheral nerve fibres, neuropeptides like substance P, calcitonin gene-related peptide, NGF, NGF-R, PGP 9.5 neuronal marker and TRPV1 as well as inflammatory/structural changes. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Odontology, Section of Oral Medicine, Clinical Oral Physiology, Oral Pathology & Anatomy, Copenhagen, Denmark